CLINICAL TRIAL: NCT01938781
Title: Optimized Treatment and Regression of HBV-induced Liver Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking University People's Hospital (Other); RenJi Hospital (Other); Peking University (Other); Shanghai Zhongshan Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Public Health Clinical Center (Other Government); Nanfang Hospital, Southern Medical University (Other); Sir Run Run Shaw Hospital (Other); Beijing YouAn Hospital (Other); Peking University First Hospital (Other); Beijing 302 Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Ditan Hospital (Other); Beijing Tiantan Hospital (Other); Huashan Hospital (Other); Tongji Hospital (Other); Tang-Du Hospital (Other); Fifth Hospital of Shijiazhuang City (Other); Logistics University of Chinese People's Armed Police Forces (Other); The First Affiliated Hospital of Shanxi Medical University (Other); The Affiliated Hospital of Yanbian University (Other)
Responsible Party: Principal Investigator, Hong You, Vice-Director of Liver Research Center, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013ZX10002004-1
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Liver Fibrosis
Keywords: Hepatitis B; Liver fibrosis; Regression; Efficacy
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B | interventions — entecavir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entecavir monotherapy (Active Comparator): entecavir, 0.5mg, qd, oral, for 2 years.
  Interventions: Drug: entecavir
- Entecavir plus peg-IFN Therapy (Experimental): entecavir combined peg-IFN in the middle 1 year.
  Interventions: Drug: entecavir; Drug: Peg-IFN

INTERVENTIONS:
Drug: entecavir — antiviral therapy
  Other Names: entecavir dispersible tablets
Drug: Peg-IFN — antiviral and antifibrosis therapy
  Other Names: Pegasys
  Arms: Entecavir plus peg-IFN Therapy

SUMMARY:
Patients with chronic hepatitis B histologically confirmed of liver fibrosis S2/S3 (similar to metavir F2/F3, Ishak 2/3/4) are randomly assigned in a 1:1 ratio. One arm is entecavir alone for 2 years; the other is entecavir alone for the first 0.5 year, entecavir plus pegylated interferon (peg-IFN) for 1 year, entecavir for another additional 0.5 year. Patients will be assessed at baseline, at every six months for blood count, liver function test, HBVDNA, AFP, prothrombin time, thyroid function, liver ultrasonography, and Fibroscan. The second liver biopsy will be performed to evaluate regression rate of liver fibrosis 1.5 years after initial therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ages from 18 to 65 years old;
2. Male or female;
3. Treatment-naive patients with chronic HBV-induced fibrosis S2/S3 (similar to F2/F3, Ishak 2/3/4), who consent to undergo liver biopsy before and after treatment;
4. Patients with HBeAg-positive, HBVDNA>2×10<4> IU/ml or with HBeAg-negative, HBVDNA>2×10<3> IU/ml;
5. Agree to be follow-up regularly;
6. signature of written inform consent.

Exclusion Criteria:

1. Patients with decompensated cirrhosis: including ascites, hepatic encephalopathy, esophageal varices bleeding or other complications of decompensated cirrhosis or hepatocelluar carcinoma;
2. Patients who are allergic to entecavir, interferon, or their components, and those considered not suitable for medications used in this study;
3. Patients coinfection with HCV or HIV, alcoholic liver disease, autoimmune liver disease, genetic liver disease, drug-induced liver injury, severe non-alcoholic fatty liver disease or other chronic liver diseases;
4. Patients with baseline AFP level higher than 100 ng/ml and possible malignant lesion on image, or AFP level higher than 100 ng/ml for continuous three months;
5. Creatinine >1.5×ULN;
6. Patients with other uncured malignant tumors;
7. Patients with severe diseases of heart, lung, kidney, brain, blood system or other organs;
8. Patients with severe neurological or psychological disease (e.g. epilepsy, depression, mania and schizophrenia);
9. Patients with poorly controlled diabetes, hypertension or thyroid disease;
10. Patients with any other reasons not suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Regression Rate of HBV-induced Liver Fibrosis | 1.5 to 2 years
  Fibrosis regression of 1 point by Ishak scoring system

SECONDARY OUTCOMES:
HBVDNA undetectable rate | 1 year and 2 years
  The HBVDNA undetectable rate after 1 year and 2-year treatment
Fibroscan scores | 1 year and 2 years
  Fibroscan scores after 1 and 2-year treatment
Life Quality | 1 year and 2 years
  Life quality after 1 and 2-year treatment by SF-36 and EQ-5D questionaire
Incidence of drug resistance | 1 year and 2 years
  Incidence of drug resistance after 1 and 2-year treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hong You, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (21):
- China (21):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - 302 Military Hospital Of China, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking Uiversity, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shijiazhuang Fifth Hospital, Shijiazhuang, Hebei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science ＆Technology, Wuhan, Hubei
  - The Affiliated Hospital of Yanbian University, Yanji, Jilin
  - Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality
  - Huashan Hospital FuDan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Hospital Affiliated to Logistics University of Chinese People's Armed Police Force, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Lu Z, Sun YM, Chen S, Meng T, Wang B, Zhou J, Wu X, Zhao X, Ou X, Kong YY, Jia J, Zhao X, You H. Multiple Low-Level Viraemia Suggest Hindered Liver Fibrosis Regression in Chronic Hepatitis B Patients During Antiviral Therapy. J Viral Hepat. 2024 Dec;31(12):898-902. doi: 10.1111/jvh.14012. Epub 2024 Oct 7. PMID 39373164